CLINICAL TRIAL: NCT03459885
Title: Long-term Paired Associative Stimulation for Rehabilitation of Lower Extremities in Persons With Incomplete Tetraplegia
Brief Title: PAS for Lower Extremity Rehabilitation in Tetraplegic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Validia Rehabilitation Centre (Unknown)
Responsible Party: Principal Investigator, Anastasia Shulga, Principal Investigator, Helsinki University Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAK 1022001
Record Dates: First submitted 2018-03-03; First posted 2018-03-09 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries; Spinal Cord Diseases
MeSH Terms: conditions — Spinal Cord Injuries; Spinal Cord Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PAS (Experimental): The intervention is given to peripheral nerve - motor cortex pairs selected by the investigator.
  Interventions: Device: Paired associative stimulation (with eXimia magnetic stimulator and Dantec Keypoint® electroneuromyography device)

INTERVENTIONS:
Device: Paired associative stimulation (with eXimia magnetic stimulator and Dantec Keypoint® electroneuromyography device) — Paired associative stimulation (PAS) administered several times per week for 8 weeks to lower limbs. PAS comprises transcranial magnetic stimulation (eXimia magnetic stimulator, Nexstim Ltd, Helsinki, Finland) and peripheral nerve stimulation (given with Dantec Keypoint® electroneuromyography device (Natus Medical Incorporated, Pleasanton, CA, USA)).

SUMMARY:
The investigators have recently shown in incomplete SCI patients that long-term paired associative stimulation is capable of restoring voluntary control over some paralyzed muscles and enhancing motor output in the weak muscles (1,2). In this study, the investigators will administer long-term paired associative stimulation to patients with incomplete cervical level SCI and investigate its effectiveness for lower extremity rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* cervical incomplete SCI

Exclusion Criteria:

* epilepsy
* metal inclusion in the head area
* pacemaker
* hearing device
* high intracranial pressure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

PRIMARY OUTCOMES:
Daniels and Worthingham's Muscle Testing | 2 days after the last stimulation session
  Leg muscle stenght is evaluated on 0-5 scale (0=no movement, 5=normal)
Daniels and Worthingham's Muscle Testing | 1 month after the last stimulation session
  leg muscles are evaluated on 0-5 scale

CONTACTS AND LOCATIONS:
Locations (1):
- BioMag laboratory, Helsinki University Central Hospital, Helsinki, Uusimaa, Finland

REFERENCES:
- [Background] Shulga A, Lioumis P, Zubareva A, Brandstack N, Kuusela L, Kirveskari E, Savolainen S, Ylinen A, Makela JP. Long-term paired associative stimulation can restore voluntary control over paralyzed muscles in incomplete chronic spinal cord injury patients. Spinal Cord Ser Cases. 2016 Jul 14;2:16016. doi: 10.1038/scsandc.2016.16. eCollection 2016. PMID 28053760
- [Background] Tolmacheva A, Savolainen S, Kirveskari E, Lioumis P, Kuusela L, Brandstack N, Ylinen A, Makela JP, Shulga A. Long-Term Paired Associative Stimulation Enhances Motor Output of the Tetraplegic Hand. J Neurotrauma. 2017 Sep 15;34(18):2668-2674. doi: 10.1089/neu.2017.4996. Epub 2017 Jul 21. PMID 28635523
- [Result] Rodionov A, Savolainen S, Kirveskari E, Makela JP, Shulga A. Effects of Long-Term Paired Associative Stimulation on Strength of Leg Muscles and Walking in Chronic Tetraplegia: A Proof-of-Concept Pilot Study. Front Neurol. 2020 May 20;11:397. doi: 10.3389/fneur.2020.00397. eCollection 2020. PMID 32508738